Skin Care Network 3 Church Passage Wood Street Barnet EN5 4QS



## **Patient Consent Form**

| Short Title | IRAS 240419 |
|---|---|
| Title | Efficiency of Presurgical Basal Cell Carcinoma margin mapping using Optical Coherence Tomography |
| Protocol Number | IRAS 240419 Protocol V04 |
| Project Sponsor | Michelson Diagnostics Ltd |
| Principal Investigator | Dr Howard Stevens |
| Patient Identification Number for this trial: | |
| Patient Clinic Identification Number: | |
| Declaration by Participant (Please initial each box) | |
| 1. I have read | the Participant Information Sheet. |
| 2. I understar<br>the project | nd the purposes, procedures and risks of the research described in . |
| laboratorie<br>Network co | mission for my doctors, other health professionals, hospitals or s outside this clinic to release information from the Skin Care oncerning my disease and treatment for the purposes of this project. In that such information will remain confidential. |
| during the where it is i | nd that relevant sections of my medical notes and data collected study may be looked at by individuals from regulatory authorities relevant to my taking part in this research. I give permission for these to have access to my records |

| 5. I have had an opportunity to ask questions and I am satisfied with the answers I have received. | |
|---|---|
| 6. I freely agree to participate in this research project as described and understand that I am free to withdraw at any time during the study without affecting my future health care. | |
| 7. I understand that I will be given a | signed copy of this document to keep. |
| Name of Participant | |
| (please print) | |
| Signature | Date |
| Name of Witness<br>(please print) | |
| Signature | Date |
| Declaration by Study Doctor/Senior Researcher <sup>†</sup> | |
| I have given a verbal explanation of the research project, its procedures, and risks and I believe that the participant has understood that explanation. | |
| Name of Study Doctor/Senior Researcher <sup>†</sup> (please print) | |
| Signature | Date |
| 1 | l l |